CLINICAL TRIAL: NCT01163500
Title: Coenzyme Q10 in Relation of the Lipid Peroxidation, Antioxidant Enzyme Activities in Coronary Artery Disease Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S07240
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pill (Placebo Comparator)
  Interventions: Other: Placebo
- Coenzyme Q10 (Experimental)
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — coenzyme Q10 supplements 60 mg/day and 150 mg/day
  Arms: Coenzyme Q10
Other: Placebo — Placebo controlled (dextrin)
  Arms: Pill

SUMMARY:
Coenzyme Q10 (Ubiquinone) is recognized as an endogenous fat-soluble antioxidant in the mitochondrial membrane and considered as a preventive factor for coronary artery disease (CAD). However, the relationships between coenzyme Q10 and the prevention of the risk of CAD are still inconsistent. The purposes of this study are to investigate the relation of coenzyme Q10 concentration with the blood lipid levels, plasma homocysteine, the markers of lipid peroxidation (TBARS, ox-LDL),antioxidant enzymes activities (catalase, glutathione peroxidase, superoxide dismutase)and to examine the association with the risk of CAD.The CAD patients is identified by cardiac catheterization as having at least 50% stenosis of one major coronary artery (n = 100). The second year is a double-blind, placebo-controlled intervention study. CAD subjects (n = 60) are randomly assign to one of the three groups (coenzyme Q10 supplements 60 mg/d, 150 mg/d, and placebo groups, n = 20/group). Intervention is going to administration for three months. The third year is a case-control study. The control group （n = 100） is comprised of healthy individuals with normal blood biochemical values, and match by age and gender with the first year CAD subjects (case group). Fasting blood samples will be obtain to determine the concentration of coenzyme Q10, homocysteine, the markers of lipid peroxidation,antioxidant enzymes activities. The differences between case and control groups will be compared by using Student's t-test. Conditional logistical regression model will be performed to calculate the odds ratio for CAD based on coenzyme Q10 level. Hopefully, the results of this study could provide the information to what has been know in CAD subjects. We expect coenzyme Q10 could be a preventive supplement to reduce the risk of CAD.

ELIGIBILITY:
Inclusion Criteria:

* CAD patients is identified by cardiac catheterization as having at least 50% stenosis of one major coronary artery

Exclusion Criteria:

* age < 18 years old
* pregnancy women
* taking lowering lipid drug (Statin)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Reducing lipid peroxidation and increasing antioxidant enzyme activities | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan